CLINICAL TRIAL: NCT06806800
Title: Venous Thromboembolism During the COVID-19 Pandemic: Evaluation of the Association With the Vaccine and COVID-19 Infection
Brief Title: Venous Thromboembolism During COVID-19 Pandemic: Evaluation of the Association With the Vaccine and COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: TEVAC-19
Record Dates: First submitted 2024-11-28; First posted 2025-02-04 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-11

CONDITIONS: Venous Thromboembolism
Keywords: TVP
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational, spontaneous, retrospective, multicenter national study for adult patients, not hospitalized, attending the Thrombo-Embolic Emergency Clinic of the Angiology and Coagulation Disorders Unit (SSD Angiologia e Malattie della Coagulazione) at the IRCCS Azienda Ospedaliero-Universitaria di Bologna, from 01/01/2018 to 31/03/2022, in whom venous thromboembolic events were suspected or confirmation was requested, as they were previously seen at another facility and referred to the reference center SSD Angiologia e Malattie della Coagulazione.

To achieve the primary objective, a case-control study will be conducted by cross-referencing data from the outpatient records of the SSD Angiologia e Malattie della Coagulazione from 29/02/2020 to 31/03/2022 with data related to SARS-CoV-2 infections provided by the Public Health Department of the Bologna Local Health Authority (Azienda USL di Bologna).

Additionally, data from the outpatient records of the SSD Angiologia e Malattie della Coagulazione from 27/12/2020 to 31/03/2022 will be integrated with data on vaccination status, date of administration, and type of vaccine administered, also provided by the Public Health Department of the Bologna Local Health Authority.

To achieve the secondary objective, data from the outpatient records of the SSD Angiologia e Malattie della Coagulazione from 01/01/2018 to 28/02/2020 will be used to describe the patient population attending the clinic during the COVID-19-free period, and will be compared with data from the period 29/02/2020 to 31/03/2022, which corresponds to the COVID-19 period.

DETAILED DESCRIPTION:
There are numerous studies exploring the epidemiology and pathophysiology of hypercoagulability associated with Sars-CoV-2 infection, while research is still ongoing to understand the relationship between thromboembolic events and the Covid-19 vaccination. With this study, the investigators aim to confirm the data already present in the literature and examine the association between thromboembolic events and infection or vaccination, focusing on the population residing in the area of the Azienda USL of Bologna.

The study is observational, retrospective, multicenter, and spontaneous, involving adult, non-hospitalized patients attending the Urgent Thromboembolic Care Clinic of the SSD Angiology and Coagulation Diseases at the IRCCS Azienda Ospedaliero-Universitaria of Bologna, from January 1, 2018, to March 31, 2022. Patients are referred to the center for suspected or confirmed venous thromboembolic events after being seen in other facilities. Treatment is provided according to clinical practice, considering the physician's judgment and the information contained in the Technical Sheet of each drug used.

The main objective of the study is achieved through a case-control study, cross-referencing the data from the outpatient reports of the SSD Angiology and Coagulation Diseases (from February 29, 2020, to March 31, 2022) with those related to Sars-CoV-2 infections provided by the Public Health Department of the Azienda USL of Bologna. Additionally, the data on patients' vaccination status, the type of vaccine, and the date of administration (from December 27, 2020, to March 31, 2022) will be integrated.

To reach the secondary objective, the outpatient reports from the pre-Covid period (from January 1, 2018, to February 28, 2020) will be compared with those from the subsequent period (February 29, 2020 - March 31, 2022), which corresponds to the pandemic period. Patients included in the study are those who accessed the Urgent Thromboembolic Care Clinic of the SSD Angiology and Coagulation Diseases, where a venous thromboembolic event was suspected or confirmed. Each patient is followed according to standard care practices, and three distinct periods are analyzed: 1) Covid-19-free period, 2) Covid-19 period, 3) Vaccination period.

The risk factors considered in the study are: Sars-CoV-2 infection confirmed by molecular swab in the 6 months prior to the onset of symptoms (Covid-19 period) and receiving at least one dose of one of the five Covid-19 vaccines authorized in Italy in the 30 days before symptom onset (Vaccination period). Data related to both risk factors are collected from computerized archives provided by the Public Health Department of the Azienda USL of Bologna and linked to patients using the unique identifier of the tax code.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Suspected or requested confirmation of a venous thromboembolic event, as the patient was previously evaluated at another facility and referred to the SSD Angiology and Coagulation Disorders reference center
* Ability to provide informed consent

Exclusion Criteria:

* Use of anticoagulants for more than 72 hours prior to presenting at the Thrombo-Embolic Emergency Clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients attending the SSD at the IRCCS Azienda Ospedaliero-Universitaria of Bologna from 01/01/2018 to 31/03/2022 will be evaluated. Each patient was managed according to routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Venous thrombotic events and SARS-CoV-2 infection | Six months prior to enrollment
  The primary objective is to identify venous thrombotic events in patients who have had prior SARS-CoV-2 infection within the previous six months
Venous thrombotic events and anti-SARS-CoV-2 vaccine | 30 days from SARS-CoV-2 vaccine administration
  The primary objective is to identify venous thrombotic events in patients who have developed symptoms within 30 days of SARS-CoV-2 vaccine administration

CONTACTS AND LOCATIONS:
Overall Officials: Benilde Cosmi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azianda Ospedaliero-Universitaria di Bologna, Bologna, Italy